CLINICAL TRIAL: NCT01419301
Title: Mindfulness Based Stress Reduction in MS
Brief Title: Mindfulness Based Stress Reduction in Multiple Sclerosis (MS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Principal Investigator, Lauren Krupp, Professor, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Teva186557-1
Record Dates: First submitted 2010-11-05; First posted 2011-08-18 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; glatiramer acetate; stress reduction; medication adherence
MeSH Terms: conditions — Multiple Sclerosis; Medication Adherence | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Mindfulness based stress reduction (MBSR) — Mindfulness based stress reduction (MBSR) is program based on daily meditation practice that guides an individual towards increased awareness and self-regulation of thoughts and actions. MBSR is easier to implement and may be shown to be more effective than cognitive-behavioral stress reduction, and is more applicable to patients with chronic illness.

SUMMARY:
This study focuses on stress, cognition, mood and fatigue and its effect on medication compliance. Medication compliance is measured by the weight of discarded needles. The investigators will be administering neuropsychological testing at baseline and the final visit. The subjects will complete self-report assessments during their 8 weeks in the study.

Group A will have additional weekly phone support for meditation, while Group B will have meditation training only.

ELIGIBILITY:
Inclusion Criteria:

* Patients with either definite MS according to the revised McDonald criteria (Polman 2005) or patients with CIS (defined as an initial MS relapse with objective documentation and 2 or more lesions within the CNS of which at least one must involve the brain)
* Patients on GA therapy for at least 6 months
* Age 18 - 70

Exclusion Criteria:

* Unwilling to comply with study procedures
* Use of other DMT in conjunction with GA
* Unable to provide informed consent.
* Current (past 30 days) substance abuse
* Newly initiated (past 30 days) psychiatry treatment
* Enrolled in another program of meditation in the past six months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-05; Primary Completion 2013-04 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Electronic measure of needle disposals (MEMS TrackCaps) | Medication adherence will be measured by total number of missed doses, calculated from total needle disposals. The total number of missed doses across the six weeks will be compared between the two treatment groups at study end.
  During the six-week MSBR program, medication adherence will be monitored with a widely used electronic measure of needle disposals (MEMS TrackCaps) This method has been demonstrated to be more accurate in MS than data obtained from either self-report or interview. At one month intervals the patient will bring the needle container to the Study Coordinator. All patients who attend at least introduction session and one telephone session will be included in the analysis.

SECONDARY OUTCOMES:
Perceived Stress Scale-10 | Baseline, 1 X between weeks 3-7, Week 8
  A 10-item scale of global perceived stress, where each item is rated from 1 to 5 according to intensity of stressor.
Holmes and Rahe Social Readjustment Rating Scale (SRRS | Baseline, 1 X between weeks 3-7, Week 8
  Stressful life events will be rated using the SRRS, which asks subjects to check if they have experienced any of a series of life events. We will use a modification of the scale used in previous MS research that eliminates several items specifically associated with MS disease activity (e.g., "major illness or injury", "sexual difficulties", "pregnancy"). The SRRS differentiates three types of stress: positive ("outstanding personal achievement"), major negative stress (death of family member), conflict and disruption in routine (e.g., family or job conflict, life changes).
Chicago Multiscale Depression Inventory (CMDI) | Baseline, 1 X betweeen Weeks 3-7, Week 8
  CMDI is a self-report questionnaire designed specifically for use in MS and other medical patient groups. It has vegetative, mood, and evaluative scales consisting of 14 items each. The use of the CMDI makes it possible to separate out neurovegetative symptoms of depression which are a potential confound in medical populations such as MS
State Trait Anxiety Inventory (STAI) | Baseline, 1 X betweeen Weeks 3-7, Week 8
  The STAI is a widely used measure of state and trait anxiety. We will focus on the measurement of state related anxiety in this study.
Positive and Negative Affect Scale (PANAS) | Baseline, 1 X between Weeks 3 - 7, Week 8
  ; Watson, Clark & Tellegen, 1989): State related positive and negative affect will be assessed by the well validated PANAS scales.
Fatigue Severity Scale (FSS) | Baseline, 1 X between Weeks 3 - 7, Week 8
  The fatigue severity scale is a reliable and valid commonly used measure of the frequent symptom of fatigue in MS.
MACFIMS neuropsychological battery | Baseline and Week 8
  At baseline and study end, an abbreviated version of the MACFIMS will be administered. This is a standard neurocognitive battery used with studies of MS subjects and includes the SDMT, PASAT, SRT, BVMT, and 9-hole peg test.
Expanded Disability Status Scale (EDSS) | Baseline and Week 8
  Expanded Disability Status Scale is the oldest and probably the most widely utilized assessment instruments in MS for determination of neurological impairment in MS. It is the standard for characterization of MS patients and for outcomes of clinical trials. It will be used to characterize patients' level of disability.
Physiologic Markers of Stress | Baseline and Week 8
  DHEA, epinephrine, and norepinephrine.
Physiologic Maker of Stress | Baseline, 1 X between Week 3 - 7, Weeek 8
  cortisol

CONTACTS AND LOCATIONS:
Overall Officials: Lauren B Krupp, M.D., Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University, Stony Brook, New York, United States